CLINICAL TRIAL: NCT04488718
Title: Evaluation of Tolerance and Acceptability of EnergieShake® Junior Powder Complete
Brief Title: ESj- Powder Complete T&A Study
Acronym: ESj
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anaiah Healthcare Pvt Ltd (Industry)
Collaborators: Brighton and Sussex University Hospitals NHS Trust (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESj-01
Record Dates: First submitted 2020-07-20; First posted 2020-07-28 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Child Nutrition Disorders; Child Malnutrition
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EnergieShake® Junior Powder Complete (test) (Experimental): EnergieShake® Junior Powder Complete will be consumed by children, as a supplement to normal diet, over a period of 7 day period to determine its acceptability (liking, compliance) and tolerance (gastro-intestinal tolerance). The dose will be the same as currently consumed product (all children recruited to the study will be consuming an oral nutritional supplement).
  Interventions: Other: EnergieShake® Junior Powder Complete

INTERVENTIONS:
Other: EnergieShake® Junior Powder Complete — Oral Nutritional Supplement

SUMMARY:
The goal of this study is to gather data on the tolerance and acceptability of a new ONS (ESj-powder complete) in children currently taking ONS.

DETAILED DESCRIPTION:
The goal of this study is to demonstrate the tolerance and acceptability of the test product when consumed by children who are currently prescribed (a similar) ONS. The data generated from this study will be submitted to the ACBS, who will consider it for reimbursement as a Food for Special Medical Purpose (FSMP) in the UK.

ELIGIBILITY:
Inclusion Criteria:

* >1-18 years of age
* Children currently prescribed and consuming Oral Nutritional Supplements (ONS)
* Willingness to take part in the study, and consent to the study protocol signed by parent/guardian or older child (when appropriate)

Exclusion Criteria:

Participants requiring exclusive enteral tube feeding

* Participants on parenteral nutrition
* Participants with cow's milk or soy allergy or lactose intolerance
* Participants with galactosaemia
* Participants with a chronic renal or liver disease
* Participants who are acutely unwell

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-04-24 (Estimated); Study Completion 2021-05-24 (Estimated)

PRIMARY OUTCOMES:
Acceptability & Tolerance: questionnaire | 7 days
  Acceptability of test product will be tested in children using a questionnaire with a liking scale (Liking Scale - 1-10 - 0 being dislike and 10 being like a lot) and compliance (intake/day versus prescribed dose) of the test product over a 7 day period and compared to acceptability when consuming their current oral nutritional supplement
Gastrointestinal Tolerance | 7 days
  Gastrointestinal (GI) tolerance of test product will be determined in children using a questionnaire detailing daily bowel habits and symptoms that occur (new or worsening) while consuming the test product over a 7 day period and compared to GI tolerance when consuming their current oral nutritional supplement. This is established using a combination of the Bristol Stool Chart scoring (BSC - type 1 up to type 7) before and during the study along with number of bowel movements/day and stool consistency.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Brighton & Sussex NHS Trust, Brighton
  - Leeds Children's Hospital,, Leeds
  - Great Ormond Street Hospital Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No
no plan